CLINICAL TRIAL: NCT01579253
Title: Untersuchungen Zur Verlaufskontrolle Bei Re-Bestrahlung Von Glioblastompatienten Mittels Kombinierter [18F]FET-PET-Kernspintomographie
Brief Title: Combined O-(2-[18F]Fluoroethyl)-L-tyrosine (FET) Positron Emission Tomography (PET) and Simultaneous Magnetic Resonance Imaging (MRI) Follow-up in Re-irradiated Recurrent Glioblastoma Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Ludwig-Maximilians - University of Munich (Other)
Responsible Party: Principal Investigator, Dr. med. Dipl.-Phys. Maximilian Niyazi, Principal Investigator, Ludwig-Maximilians - University of Munich
Other Study IDs: 361-11
Record Dates: First submitted 2012-04-15; First posted 2012-04-17 (Estimated); Last update posted 2012-12-18 (Estimated); Status verified 2012-12

CONDITIONS: Glioblastoma; Nervous System Neoplasms; Central Nervous System Neoplasms; Astrocytoma; Glioma; Neoplasms, Neuroepithelial; Neuroectodermal Tumors; Neoplasms by Histologic Type; Neoplasms, Nerve Tissue
Keywords: Recurrent glioblastoma; Radiotherapy; PET-MRI; FET-PET
MeSH Terms: conditions — Glioblastoma; Nervous System Neoplasms; Central Nervous System Neoplasms; Astrocytoma; Glioma; Neoplasms, Neuroepithelial; Neuroectodermal Tumors; Neoplasms by Histologic Type; Neoplasms, Nerve Tissue

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Patients with recurrent glioblastoma who are planned to receive a second course of radiation are to be included into this monocentric cohort trial. Due to multiple pre-treatments simultaneous combined positron emission tomography (PET) with O-(2-[18F]fluoroethyl)-l-tyrosine (FET) as well as magnetic resonance imaging (MRI) is used for treatment planning and follow-up imaging as it allows for a better distinction between treatment-related changes and viable tumor tissue.

DETAILED DESCRIPTION:
For glioblastoma (GBM) patients it has been proven that a [18F]FET-PET scan is very helpful especially in target volume definition and after the treatment, in turn, the combination of MRI and [18F]FET-PET is diagnostically most useful to distinguish between radiation necrosis and a real progressive disease.

The response to therapy is based on the newly formulated Revised Assessment in Neuro-Oncology (RANO) criteria. Kinetic and static [18F]FET-PET scans are useful to supplement this modality and its own prognostic value concerning relapsing patients will be examined.

The special feature of this study is the use of both modalities in parallel, allowing simultaneous acquisition of morphological changes, functional and molecular imaging.

Secondary methodological issues are dealt with, such as the relationship between contrast uptake, perfusion and [18F]FET uptake. In this regard, the hybrid imaging may serve for hypothesis generation, as in parallel in a unique way of contrast enhancement and tracer kinetics can be investigated (simultaneous contrast-enhanced analysis and tracer application).

In particular, FET kinetics are examined in more detail (for example, differences between increasing and decreasing kinetics) to find ways of how to use certain MRI sequences for better visualization of viable tumor tissue and vice versa .

ELIGIBILITY:
Inclusion Criteria:

* 18 - 75 years old
* histologically or magnetic resonance imaging proven recurrent glioblastoma
* re-irradiation possible
* willing and able to give free informed consent

Exclusion Criteria:

* not willing or able to give free informed consent
* pregnancy
* claustrophobia
* metallic objects or implanted medical devices in the body

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with recurrent glioblastoma who are planned to receive a re-irradiation
Sampling Method: Non-Probability Sample
Enrollment: 10 (Estimated)
Dates: Start 2012-04

CONTACTS AND LOCATIONS:
Overall Officials: Maximilian Niyazi, MD, MSc, Principal Investigator — Ludwig-Maximilians - University of Munich
Locations (1):
- University of Munich, Dep. of Radiation Oncology, Munich, Bavaria, Germany